CLINICAL TRIAL: NCT03718338
Title: Mechanisms of Metabolic and Hormone Action on Plaque Formation in Brain and Carotid Vessels in Men Undergoing Androgen Deprivation Therapy
Brief Title: Mechanisms of Metabolic and Hormone Action on Plaque Formation in Brain and Carotid Vessels in Patients With Prostate Adenocarcinoma
Status: Terminated | Type: Observational
Why Stopped: Terminated due to low accrual
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RG1001903; 9939 (Other: FHCRC); NCI-2018-01618 (Registry Identifier: CTRP); 5P30CA015704 (NIH)
Record Dates: First submitted 2018-09-12; First posted 2018-10-24 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical Evaluations: Patients undergo clinical evaluations over 12 months including physical exam and vital signs, waist to hip circumference, medical history and events, laboratory evaluations, imaging evaluations, cognitive function evaluations, gait assessment, and quality of life questionnaires.
  Interventions: Procedure: Evaluation; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Evaluation — Undergo clinical evaluations
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This trial studies the mechanisms of metabolic and hormone action on plaque formation in brain and carotid vessels in patients with prostate adenocarcinoma. Studying the biomarkers in the laboratory may help doctors know the impact of androgen deprivation on metabolic, brain and cardiovascular endpoints.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo clinical evaluations over 12 months including physical exam and vital signs, waist to hip circumference, medical history and events, laboratory evaluations, imaging evaluations, cognitive function evaluations, gait assessment, and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically confirmed adenocarcinoma of the prostate
* Non-castrate disease with a serum testosterone level >= 50 ng/dL (1.73 nmol/L) at baseline
* No evidence of distant metastatic disease on baseline computed tomography-chest, abdomen and pelvis (CT-CAP) and bone scans
* Patients will be stratified by the presence or absence of pre-existing cardiovascular disease defined as at least one of the following:

  * Prior myocardial infarction >= 30 days before enrollment
  * Prior revascularization procedure >= 30 days before consent, including:

    * Coronary artery stent placement or balloon angioplasty
    * Coronary artery bypass graft surgery
    * Stent placement or balloon angioplasty to a carotid, iliac, femoral, or popliteal artery
    * Carotid endarterectomy surgery
    * Vascular bypass surgery of the iliac, femoral, or popliteal artery
  * Results from angiogram or CT angiogram of coronary, carotic, iliac, femoral, or popliteal arteries that documents at least one vascular stenosis >= 50% at any time point before enrollment
  * Carotid ultrasound results that shows stenosis >= 50% at any time point before enrollment
  * Ankle-brachial pressure index < 0.9 at any time point before enrollment
* Intent to initiate continuous androgen deprivation therapy (ADT) for at least 12 months

Exclusion Criteria:

* No prior treatment with ADT at time of study entry. (Prior neoadjuvant/adjuvant ADT is allowed only if the last injection of a depot formulation wore off at least 12 months prior to enrollment)
* Previous or concurrent hormonal or systemic therapy for prostate cancer including: anti-androgens, estrogens, megestrol acetate, ketoconazole, abiraterone, enzalutamide, or chemotherapy. (Prior or planned neoadjuvant bicalutamide for prevention of tumor flare is allowed)
* Plans to start or continue treatment with an investigational product after enrollment
* Poorly controlled type 1 or type 2 diabetes mellitus, based on hemoglobin A1c, as judged by the investigator
* Prior or planned surgical castration
* Poorly controlled hypertension at time of study entry, as judged by the investigator
* Myocardial infarction or stroke < 30 days prior to enrollment
* Coronary, carotid, or peripheral artery revascularization < 30 days prior to enrollment
* Planned or scheduled cardiac surgery or percutaneous coronary intervention (PCI) procedure that is known at the time of enrollment
* Mental incapacity or language barrier precluding adequate understanding or cooperation
* Inability to tolerate magnetic resonance imaging (MRI) imaging, or both Lupron and Degarelix
* Any other clinically significant disorder which may affect the subject's health or the outcome of the trial as judged by the investigator
* Estimated glomerular filtration rate (eGFR) < 45
* History of allergy to gadolinium contrast agent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with prostate adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change in visual characterization of 18F-florbetapir (Amyvid) positron emission tomography (PET) scans results after Andorgen Deprivation Therapy | 12 Months
  Change From Baseline visual characterization scan results at 12 months
Change standardized uptake values of 18F-florbetapir (Amyvid) positron emission tomography (PET) scans results | 12 Months
  Change from baseline standardized uptake values in select regions of interest at 12 months

SECONDARY OUTCOMES:
Cognitive test results: Story recall | 12 months
  Change in baseline Story Recall results at 12 months
Cognitive Test Results: Change in Montreal Cognitive Assessment (MOCA) | 12 Months
  Change in baseline MOCA score results at 12 months
Cognitive Test Results: Change in Clinical Dementia Rating Scale | 12 Months
  Change in baseline Clinical Dementia Rating Scale score at 12 months
Cognitive Test Results: Digit span | 12 Months
  Change in baseline Digit span results at 12 months
Cognitive Test Results: Letter number sequencing | 12 Months
  Change in baseline Letter number sequencing results at 12 months
Cognitive Test Results: Stroop Test Results | 12 Months
  Change in baseline Stroop Test Results at 12 months
Cognitive Test Results: Symbol Digit Modalities Test | 12 Months
  Change in baseline Symbol Digit Modalities Test score at 12 months
Cognitive Test Results: Visuo-Spatial Learning Test | 12 Months
  Change in baseline Visuo-Spatial Learning Test results at 12 months
Cognitive Test Results: Rey auditory verbal learning test (RVLT) | 12 Months
  Change in baseline Rey auditory verbal learning test (RVLT) score at 12 months
Inflammatory and immune markers: Change in CRP | 12 Months
  Change in baseline CRP values at 12 months
Inflammatory and immune markers: Change in IGFBP3 | 12 Months
  Change in baseline IGFBP3 at 12 months
Inflammatory and immune markers: Change in IGFBP1 | 12 Months
  Change in baseline IGFBP1 at 12 months
Inflammatory and immune markers: Change in IGF-1 | 12 Months
  Change in baseline IGF-1 at 12 months
Inflammatory and immune markers: Change in IL-6 | 12 Months
  Change in baseline IL-6 at 12 months
Metabolic Markers: Change in HgbA1C | 12 Months
  Change in baseline HgbA1C at 12 months
Metabolic Markers: Change in Estradiol | 12 Months
  Change in baseline Estradiol at 12 months
Metabolic Markers: Change in Follicle Stimulating Hormone (FSH) | 12 Months
  Change in baseline Change in Follicle Stimulating Hormone (FSH) at 12 months
Metabolic Markers: Change in Leptin | 12 Months
  Change in baseline Leptin at 12 months
Metabolic Markers: Change in Adiponectin | 12 Months
  Change in baseline Adiponectin at 12 months
Metabolic Markers: Change in homeostatic model assessment of insulin resistance (HOMA-IR) | 12 Months
  Change in baseline HOMA-IR values at 12 months; Calculated based on fasting glucose and insulin test results.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Yu, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No